CLINICAL TRIAL: NCT06298981
Title: Pulse Rate and Breathing Rate Accuracy Study - NuraLogix AMC-SDK
Brief Title: Pulse Rate and Breathing Rate Accuracy
Status: Recruiting | Type: Observational
Sponsor: Nuralogix Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2301
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Pulse Rate and Breathing Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: noninvasive and investigational NuraLogix AMC-SDK — The NuraLogix AMC-SDK is a noninvasive device that allows for real-time, remote measuring using facial recordings.

SUMMARY:
The purpose of this study is to conduct a Breathing Rate and Pulse Rate accuracy validation comparing the NuraLogix AMC-SDK to the Reference devices, an FDA cleared End Tidal Carbon Dioxide monitor (GE Datex-Ohmeda) and a standard ECG (GE Datex-Ohmeda) derived heart rate reference. This will be done by manually scoring the collected waveform for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have the ability to understand and provide written informed consent or have legally authorized representative consent to participate
* Participant must be 18 to 81 years of age (≥ 18 age to < 82)
* Participant must be willing and able to comply with study procedures and duration
* Participants or legally authorized representative must be able to read or write in English

Exclusion Criteria:

* Participants who refuse or are unable to provide to sign an informed written consent for study
* Participants evaluated by the Investigator and Clinical Staff and found to be medically - unsuitable or have self-reported health conditions that are currently unstable as identified in the Health Assessment Form and Health Screening
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor Region of Interest (ROI) which would limit the ability to test ROI needed for the study. Tattoo in the optical path which would limit the ability to test ROI needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the particular areas utilized.)
* Participants with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, or other medical sensors (self- reported)
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of diversity in race, age, gender, BMI, skin tone, and health conditions. The health conditions will constitute inclusion of healthy controls (to allow testing over the full range of breaths per minute) and disease comorbidities (to represent comorbidities such as COPD, CHF, Asthma, Diabetes, Hypertension, and Obesity). An attempt will be made to enroll a variety of skin tones.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Breathing rate accuracy validation | 1-2 hours
  The purpose of this study is to conduct a Breathing Rate accuracy validation comparing the NuraLogix AMC-SDK to the Reference, an FDA cleared End Tidal Carbon Dioxide monitor (GE Datex-Ohmeda) by manually scoring the collected waveform for data analysis
Pulse rate accuracy validation | 1-2 hours
  This study will also assess the pulse rate measurements of the NuraLogix AMC-SDK for comparison to a standard ECG (GE Datex-Ohmeda) derived heart rate reference.

SECONDARY OUTCOMES:
Pulse rate simulation | 1-2 hours
  To assess a broader pulse rate range by manipulating the speed of recorded videos.

CONTACTS AND LOCATIONS:
Locations (1):
- Element Materials Technology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD